CLINICAL TRIAL: NCT02773017
Title: The ED50 of DEX for Providing Sedation in Different Female Age Group
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX sedation
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Combined Spinal-epidural Anesthesia
Keywords: sedation; age; dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Youth female group (Experimental): patients in the Youth female group, aged 20~35, were accepted an initial dose of 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last three turning points.
  Interventions: Drug: Dexmedetomidine A
- Middle-aged female group (Experimental): patients in the Middle-aged female group, aged 40~60, were accepted an initial dose of 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last three turning points.
  Interventions: Drug: Dexmedetomidine B
- Elderly female group (Experimental): Patient in the elderly female group, aged 65~79, were accepted an initial dose of 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last three turning points.
  Interventions: Drug: Dexmedetomidine C

INTERVENTIONS:
Drug: Dexmedetomidine A — initial dose was 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last three turning points.
  Other Names: Dexmedetomidne in youth female group
  Arms: Youth female group
Drug: Dexmedetomidine B — initial dose was 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last three turning points.
  Other Names: Dexmedetomiodine in middle-age female group
  Arms: Middle-aged female group
Drug: Dexmedetomidine C — initial dose was 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last three turning points.
  Other Names: Dexmedetomidine in elderly female group
  Arms: Elderly female group

SUMMARY:
Dexmedetomidine(DEX) could provide dose-dependent sedation , analgesia , anti-anxiety and inhibition of sympathetic nerves and other effects. Because of its minimal impact on the respiratory , currently it was more and more widely used to sedate patients undergoing regional anesthesia.Many anesthetic pharmacokinetics and pharmacodynamics are often affected by age, and current studies with regard to the effects of age on dexmedetomidine pharmacodynamic are rare. This study was designed to explore the right DEX dose of different female Age of patients to produce suitable sedation.Dexmedetomidine be used in patients with combined spinal and epidural anesthesia for sedation,which is monitored by the Narcotrend,during the operation.The relation between Narcotrend index (NTI) and the depth of sedation for patients is also investigated.

DETAILED DESCRIPTION:
90 patients scheduled for combined spinal epidural spinal anesthesia were included in one of three groups. In each group,determination of median effective (ED50) doses was performed by the Dixon up-and-down method, an initial dose of 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1 μg/kg in first three turning points and 0.05μg/kg in the last three turning points.Initial doses was 1.4μg/kg, .Sedative efficacy was defined as an OAA/S of ≤3,30 min after the beginning of drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ patient undergoing lower extremity surgery
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18.0～25.0kg/m2

Exclusion Criteria:

1. Mental illness can not match
2. epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. People who were language or hearing impaired
5. Sensory block reached to T8 or higher.
6. People who had lung infection or sleep apnea syndrome.
7. Pregnancy
8. Chronic renal failure
9. Alcohol or drug abuse
10. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug

    -

    -

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The ED50 of DEX for providing sedation | 30min after the start of the infusion
  The aim of this study is to define the optimum bolus dose (ED50) of dexmedetomidine for producing adequate sedation during spinal anesthesia in different female age group using the Dixon and Mood up-and-down method。

SECONDARY OUTCOMES:
The ED95 of DEX | 30min after the start of the infusion
  To determine the optimum bolus dose (ED95) of dexmedetomidine for producing adequate sedation during spinal anesthesia in different female age group.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China